CLINICAL TRIAL: NCT06798675
Title: A PHASE 2A, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL GROUP, DOSE-RANGING CLINICAL TRIAL TO EVALUATE THE PHARMACOKINETICS, PHARMACODYNAMICS, AND SAFETY OF nC-001 IN PATIENTS WITH CHRONIC EUVOLEMIC HYPONATREMIA
Brief Title: Phase 2a Study for PK/PD of nC-001
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: nephCentric (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PNC-101
Record Dates: First submitted 2025-01-07; First posted 2025-01-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: CHRONIC HYPONATREMIA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 15gm (Active Comparator)
  Interventions: Drug: nC-001
- 30gm (Active Comparator)
  Interventions: Drug: nC-001
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: nC-001 — solid dosage form single dose
  Arms: 15gm; 30gm
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
CHRONIC EUVOLEMIC HYPONATREMIA

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥18 and ≤85 years of age
2. Diagnosis of chronic euvolemic hyponatremia

Exclusion Criteria:

* 1. Hyponatremia assessed by the Investigator to be hypervolemic, hypovolemic, or due to psychogenic polydipsia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Serum Urea and Sodium (Na) | 24 hrs

SECONDARY OUTCOMES:
Safety | 15 days
  Incidence and severity of treatment-emergent adverse events (TEAE) as assessed by CTCAE v5.0
Tolerability | 1 day
  Five-Point Palatability Scale; (scores 1-5)
  1. Very Bad
  2. Bad
  3. Neutral
  4. Good
  5. Very Good